CLINICAL TRIAL: NCT00855452
Title: rIL-2 Activated Allogeneic Lymphocytes for the Induction of Graft Versus Tumor Effect (GVT) in Metastatic Solid Tumors
Brief Title: Activated Allogeneic Lymphocytes for Induction Graft Versus Tumor Effect in Metastatic Solid Tumors
Acronym: rIL-2(LAK)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Prof. Reuven Or, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0457-08-HMO-CTIL
Record Dates: First submitted 2009-02-19; First posted 2009-03-04 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2008-10

CONDITIONS: Metastatic Breast Cancer; Malignant Melanoma; Renal Cell Cancer; Gastrointestinal Cancer
Keywords: GVL; rIL-2(LAK); GVHD; MST; alloCT; alloBMT
MeSH Terms: conditions — Breast Neoplasms; Melanoma; Carcinoma, Renal Cell; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: one - three cycles of cell therapy during 4-6 weeks (3-5x10^7 cells/kg will be given through IV systemically — Patients will be eligible to participate in a treatment program based on systemic administration of mismatched lymphocytes activated in vitro with rIL-2(LAK) followed by rIL-2 inoculation in vivo

SUMMARY:
The present protocol is a phase 2 study designed to investigate the potential application of allogeneic cell-mediated immunotherapy in metastatic solid tumors, similarly to the well established graft versus leukemia (GVL) effects, in patients with metastatic solid tumors resistant to conventional treatment modalities. Patients will be eligible to participate in a treatment program based on systemic administration of mismatched lymphocytes activated in vitro with rIL-2 (LAK) followed by rIL-2 inoculation in vivo. This treatment is aiming to induce an anti-tumor effect mediated by the efficient killing activity of the rIL-2 activated cells. Prior to cell infusion patients will receive the conditioning treatment with low dose Cyclophosphamide (Cyc) or Fludarabine with 2 injections of low dose alpha interferon. Cell therapy will be combined with specific anti-tumor monoclonal antibodies if available for the specific disease. Further activation of the anti-tumor activity of alloreactive donor T cells and natural killer (NK) cells will be accomplished by in vivo inoculation of rIL-2, aiming for enhancing the anti-cancer potential of donor-derived effectors cells. Patients will receive one - three cycles of cell therapy, as long as there are no signs of Graft- versus - Host - disease (GVHD) and the malignant disease is controlled.

ELIGIBILITY:
Inclusion Criteria:

Consenting patients (age 12-70) will be eligible for participation in the study involving anti-tumor immunotherapy provided the following criteria are met:

1. Evidence of cancer not expected to be cured with conventional modalities:

   Pediatric patients: Chemotherapy-resistant neuroblastoma stage 4 & sarcomas. Adult patients: Metastatic breast cancer, malignant melanoma, renal cell cancer and selected cases of ovary cancer, gastrointestinal cancer, small-cell and non-small cell lung cancer with non-bulky metastatic disease, metastatic prostate cancer.
2. Patients with measurable disease evaluable for response with anticipated life expectancy >3 months.
3. Patients must be >2 weeks off anti-cancer or potentially immunosuppressive treatment.
4. Adequate ambulatory performance status (Karnofsky >80%; ECOG 0-1) to enable outpatient treatment (see Appendix 1).
5. Compliant and cooperative patients anticipated to be evaluable for response according to investigator's assessment.
6. HLA-noncompatible (partial matched or mismatched) donor available.

Exclusion Criteria:

Patients will be excluded from participation in the study if any of the following criteria are met:

1. Any of the above criteria are not met.
2. Patients with a significant history or current evidence of potentially severe cardiovascular disease.
3. Hepatic and/or renal failure.
4. Abnormal PT and PTT.
5. Patients with abnormal hemogram (PMN<1.0x109/L; HB<10; Plts<50x109/L)
6. Evidence of serious active infection requiring antibiotic therapy.
7. Evidence of active disease requiring steroid or cytotoxic therapy.
8. Pregnancy.
9. Contraindication for donation due to donor disease: HIV-1; HBsAg positivity.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
CR:disappearance of disease.PR:<50% decrease in the total tumor load of the lesions SD:<50% reduction and 25% increase in the sum of the products of the longest perpendicular diameters of the measured lesions.PD:>25% increase in the size of lesion. | on day +7 day +17, day +28 post cell therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Reuven Or, Prof., M.D., Principal Investigator — Hadassah University Hospital
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel